CLINICAL TRIAL: NCT04002986
Title: Comprehensive Genetic Assessment, Risk and Education in a Mammography Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Niloy Jewel (Jewel) Samadder, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19-004343
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Women Age 35+ Qualifies if >15% Lifetime Risk of Breast Cancer as Defined by IBIS Version 8
Keywords: increased risk of breast cancer
MeSH Terms: interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women at intermediate/high risk of breast cancer (Experimental): Women age 35 years old identified at intermediate/high risk of breast cancer will receive genetic testing
  Interventions: Genetic: Genetic Testing

INTERVENTIONS:
Genetic: Genetic Testing — A blood draw or saliva kit will be provided to collect subject cells

SUMMARY:
Researchers are trying to learn more about the prevalence of genetic mutations in women who are at intermediate/high risk of breast cancer and how that information my assist providers in improving screening and preventative options.

ELIGIBILITY:
Inclusion Criteria:

* Women participating in IRB:18-010601
* Aged 35 and over with a negative routine mammogram within 3 months.
* Qualifies as intermediate or high-risk (>15% lifetime risk of breast cancer as defined by IBIS version 8).
* Have an active email address for survey completion

Exclusion Criteria:

* Not participating in the Mayo Clinic CEDM pilot (IRB: 18-010601)
* Known genetic cancer syndrome with test results available for review in Mayo EMR
* Known breast cancer
* Unable to understand or sign informed consent

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Genetic mutations | One year
  Number of subjects to have a pathogenic/likely pathogenic mutations (Positive test result on Proactive Cancer Screening Panel)
Study Participants | One year
  Number of subjects who decide to undergo genetic panel testing

CONTACTS AND LOCATIONS:
Overall Officials: N. Jewel Samadder, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials